CLINICAL TRIAL: NCT03370757
Title: Very Low Birthweight (VLBW) Preterm Infant Skin Health With Bundled Care in the Neonatal Intensive Care Unit (NICU): A Randomized Controlled Trial
Brief Title: Very Low Birth Weight Preterm Infant Bundled Care in the NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00086595
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Preterm Infants

STUDY DESIGN:
Intervention Model Description: Infants will be randomly assigned and stratified by birth weight (≤ 800 grams, >800 grams to 1150 grams, > 1150 grams) to either 3- or 6- hour bundled diaper care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-hour bundled care (Active Comparator): Infants in this group will have their diaper changed every 3 hours during 3-hour bundled care.
  Interventions: Other: 3-hour bundled care
- 6-hour bundled care (Active Comparator): Infants in this group will have their diaper changed every 6 hours.
  Interventions: Other: 6-hour bundled care

INTERVENTIONS:
Other: 3-hour bundled care — Infants in the 3-hour bundled care group will receive diaper changes every 3 hours with observational coding, microbiome samples, skin pH measurements and trans epidermal water loss measurements taken 3 times per week.
  Arms: 3-hour bundled care
Other: 6-hour bundled care — Infants in the 6-hour bundled care group will receive diaper changes every 6 hours with observational coding, microbiome samples, skin pH measurements and trans epidermal water loss measurements taken 4 times per week.
  Arms: 6-hour bundled care

SUMMARY:
The purpose of this study is to explore the impact of bundling nursing care activities on the overall health of Very Low Birthweight (VLBW) preterm infants who receive bundled care in a Level IV Neonatal Intensive Care Unit (NICU). The study will evaluate differences in infant health when diaper changes occur at 3- versus 6-hours during 3-hour bundled care. Differences in infant skin health between 3- and 6-hour bundled care diapering at two sites (buttocks and chest) will also be evaluated.

DETAILED DESCRIPTION:
Preterm infants' growth and developmental outcomes vary with illness severity and degree of neurological insult and unpredictable variations in outcomes exist even among healthy preterm infants. The variations in preterm infants' outcomes have led to the supposition that the neonatal intensive care unit (NICU) environment may negatively impact the health and development of these infants and significant research has been devoted to examination of light, noise, and caregiving interventions. Consequently, many NICUs have implemented neuroprotective strategies to reduce over simulation, promote sleep and facilitate brain development in high-risk infants including the grouping of care activities around a single caregiving event described as "clustering" or "bundling care". Yet, the number and type of caregiving activities that are included in bundled care and the timeframe between bundled care events has not been systematically studied. The inclusion and exclusion of certain care activities in any individual care event is often dictated by the infant's treatment plan or needs, but some activities like diapering may be optional. Understanding the impact of when to include optional, yet stress provoking interventions, will allow us to minimize overall environmental stress in hospitalized very low birthweight (VLBW) infants. Therefore, given the lack of data around bundled care, the investigators aim to explore through a randomized controlled design the impact of bundling diaper care activities on overall health of VLBW preterm infants. The investigators will include a focus on skin health because it is important to understand the benefits of decreased infant stress and any potential skin health trade-offs associated with longer versus shorter time between diapering care. Findings from this study will allow us to better understand the relationship between neonatal skin health while providing developmentally appropriate bundled care.

ELIGIBILITY:
Inclusion Criteria:

1. Must be participating in the Intensive Care Nursery standard 3-hour bundled care
2. Must wear a breathable diaper
3. Must be ≤ 32 weeks gestation at birth and weigh ≤ 1500g at birth.
4. Infants are expected to remain hospitalized for at least 4 weeks

Exclusion Criteria:

1. Neonatal Abstinence Syndrome
2. Humidified incubator
3. Diaper rash
4. Pre-existing or genetic skin conditions
5. Use of barrier creams
6. Severe illness requiring 1:1 nursing care: e.g. minimal stimulation protocol, high frequency ventilation, vasopressor drug support, or body cooling.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Brandon, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brandon DH, Hatch D, Barnes A, Vance AJ, Harney J, Voigtman B, Younge N. Impact of diaper change frequency on preterm infants' vital sign stability and skin health: A RCT. Early Hum Dev. 2022 Jan;164:105510. doi: 10.1016/j.earlhumdev.2021.105510. Epub 2021 Nov 20. PMID 34896732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 2/2018 - 7/2019 Location: Level IV NICU
Pre-assignment Details: 1 infant was consented but discharged home before being randomized because the infant never reached q3 hour feedings (discharged home on G-tube).
Period: Overall Study
Arm/Group | 3-hour Bundled Care | 6-hour Bundled Care
Started | 20 | 28
Completed | 20 | 26
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3-hour Bundled Care | 6-hour Bundled Care | Total
Number analyzed (Participants) | 20 | 26 | 46
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational Age at Birth | 27.6 (2.8) | 28.4 (2.8) | 28.0 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 18 | 25
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 17 | 24 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 8 | 13 | 21
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 26 | 46

OUTCOME MEASURES:

1. Primary Outcome: Mean Heart Rate by Group
Description: Heart rate instability was defined as having a mean heart rate value during a bundled care event that was ≥1 standard deviation above or below the mean heart rate value during the 90 minutes before the event started. In addition, clinically meaningful parameters were added to indicate exceptions to this definition. For HR, mean values ≥ one standard deviation below the mean was categorized as physiologically unstable only if the mean value was < 100. Based on these criteria, each observation was categorized as physiologically unstable or not.
Time Frame: During hospitalization, approximately four weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- 3-hour Bundled Care: Infants in this group had their diaper changed every 3 hours during 3-hour bundled care.
  3-hour bundled care: Infants in the 3-hour bundled care group received diaper changes every 3 hours.
- 6-hour Bundled Care: Infants in this group had their diaper changed every 6 hours.
  6-hour bundled care: Infants in the 6-hour bundled care group received diaper changes every 6 hours.
Arm/Group | 3-hour Bundled Care | 6-hour Bundled Care
Number analyzed (Participants) | 20 | 26
beats per minute | 200 (75.19) | 185 (73.41)

2. Secondary Outcome: Estimates of Infant Buttock Transepidermal Water Loss (TEWL) by Group
Description: TEWL was measured at the beginning of each bundled care event using the DermaLab® TEWL probe (Cortex Technology, Hadsund, Denmark). Transepidermal water loss is the process of water moving through the layers of the skin and evaporating.
  Linear mixed models (LMM) were used to examine group differences in TEWL. Outcomes in these models consisted of within-subject change over time in skin TEWL of the buttock. In the model, TEWL was regressed on diaper change group and the number of days since study initiation. TEWL estimates and confidence intervals are reported by group across all bundled care observations.
Time Frame: During hospitalization, approximately four weeks
Measure: Mean (95% Confidence Interval); unit: g/m^2/h
Groups:
- 3-hour Bundled Care: Infants in this group had their diaper changed every 3 hours.
  3-hour bundled care: Infants in the 3-hour bundled care group received diaper changes every 3 hours with trans epidermal water loss measurements taken 3 times per week.
- 6-hour Bundled Care: Infants in this group had their diaper changed every 6 hours.
  6-hour bundled care: Infants in the 6-hour bundled care group received diaper changes every 6 hours with trans epidermal water loss measurements taken 4 times per week.
Arm/Group | 3-hour Bundled Care | 6-hour Bundled Care
Number analyzed (Participants) | 20 | 26
g/m^2/h | 38.48 [31.93 to 45.03] | 35.73 [29.67 to 41.79]

3. Secondary Outcome: Microbiota Diversity of the Skin at Both the Buttocks and Chest Sites and Stool by Group
Description: The Shannon Diversity index measures the alpha diversity of a bacterial sample. Function of richness and evenness of 16S rRNA gene amplicon sequence variants (i.e., proxy for prokaryote species-like groupings) within each sample. A higher Shannon diversity means that a sample had a combination of a higher number of species of archaea and bacteria, and/or a more even relative abundance of those species within a sample.
Time Frame: During hospitalization, approximately four weeks
Population: A total of 273 skin swabs from the buttocks were analyzed from infants in the 3-hr bundled care group and 255 swabs from infants in the 6-hr bundled care group. A total of 266 skin swabs from the chest were analyzed from infants in the 3-hr bundled care group and 254 swabs from infants in the 6-hr bundled care group. A total of 65 stool samples were analyzed from infants in the 3-hr bundled care group and 66 samples from infants in the 6-hr bundled care group.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Samples
Groups:
- 3-hour Bundled Care: Infants in this group had their diaper changed every 3 hours.
  Skin swabs were collected on the buttocks & chest from infants up to 3 times per week during their assigned diaper change interval from the time of initiation of the intervention until discharge. Stool samples were collected 1 time per week when available.
- 6-hour Bundled Care: Infants in this group had their diaper changed every 6 hours.
  Skin swabs were collected on the buttocks & chest from infants up to 3 times per week during their assigned diaper change interval from the time of initiation of the intervention until discharge. Stool samples were collected 1 time per week when available.
Arm/Group | 3-hour Bundled Care | 6-hour Bundled Care
Number analyzed (Participants) | 20 | 26
Number analyzed (Samples) | 604 | 575
score on a scale
  Skin-Buttocks: number analyzed (Samples) | 273 | 255
  Skin-Buttocks | 4.14 (0.67) | 3.99 (0.78)
  Skin-Chest: number analyzed (Samples) | 266 | 254
  Skin-Chest | 4.14 (0.74) | 4.18 (0.75)
  Stool: number analyzed (Samples) | 65 | 66
  Stool | 4.16 (0.70) | 3.56 (0.77)

ADVERSE EVENTS:
Time Frame: During hospitalization, approximately four weeks.
Groups:
- 3 Hour Bundled Care: Infants in this group will have their diaper changed every 3 hours during 3-hour bundled care.
- 6 Hour Bundled Care: Infants in this group will have their diaper changed every 6 hours during 3-hour bundled care.
Arm/Group | 3 Hour Bundled Care | 6 Hour Bundled Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/26
Other Adverse Events (participants affected / at risk) | 0/20 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT03370757/Prot_SAP_000.pdf